CLINICAL TRIAL: NCT00986687
Title: Oocyte Cryopreservation: A Pilot Study Comparing Fertilization and Embryo Development Between Fresh and Vitrified Sibling Oocytes
Brief Title: Oocyte Cryopreservation Comparing Fresh and Vitrified Sibling Oocytes
Status: Completed | Type: Observational
Sponsor: UConn Health (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Claudio Benadiva, Laboratory Director and Director of the Preimplantation Genetics Diagnosis Program,, UConn Health
Other Study IDs: 09-189-3; 29642
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
Keywords: Oocyte cryopreservation; vitrification
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Embryos
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vitrified oocytes
- Control oocytes

SUMMARY:
Vitrification is a method to cryopreserve biological specimens that are sensitive to chilling injury such as oocytes and embryos, and it has been employed with increased survival rate and live births (Hong et al., 1999; Kuleshova et al., 1999; Yoon et al., 2000; Chung et al 2000; Wu et al., 2001: Kuwayama et al 2006). In their study the researchers propose to directly compare oocyte survival, fertilizaton and embryo development between sibling oocytes.

The Cryotop method of vitrification, which the researchers aim to investigate in their study, has been reported as the most efficient method for human oocytes cryopreservation (Kuwayama et al, 2005, Antinori et al, 2006, Lucena et al, 2006, Cobo et al, 2008). Follow up of over 200 infants conceived from vitrified oocytes (Chian et al, 2008) indicate that the mean birth weight and the incidence of congenital anomalies are comparable to that of spontaneous conceptions in fertile women or infertile women undergoing IVF treatment.

DETAILED DESCRIPTION:
The necessity to cryopreserve human oocytes successfully, with the goal of achieving term pregnancies at rates equivalent to those obtained with fresh oocytes is urgent. Cryopreservation of oocytes is desirable because: 1) it would allow infertility patients to store excess oocytes instead of embryos, eliminating some of the ethical and religious concerns that accompany embryo storage; 2) permit storage of donor oocytes in egg banks, analogous to existing sperm banks. This option would allow the cryopreserved oocytes to be quarantined until screening for infectious diseases is completed, and would also avoid donor-recipient synchronization difficulties; and 3) can help cancer patients preserve their fertility before they face sterilization due to chemotherapy or radiation. Oocyte cryopreservation is therefore gaining in popularity as an option for infertility treatment as well as fertility preservation.

This is a pilot study to evaluate the outcomes of oocyte vitrification using the Cryotop method in women undergoing IVF, by simultaneously evaluating embryos derived from vitrified and fresh oocytes coming from the same stimulated cycle.

The primary outcome measures that will be tracked and tabulated are oocyte survival, fertilization and cleavage rate, and subsequent embryo development, compared between vitrified and fresh oocytes. Secondary outcomes are implantation, clinical pregnancy, miscarriage and live birth rates using embryos derived from the vitrified oocytes for transfer.

ELIGIBILITY:
Inclusion Criteria:

1. Females 21 to 37 years of age.
2. Normal serum follicle stimulating hormone (FSH) concentration <10 mIU/ml and estradiol (E2) concentration <70 pg/ml obtained on day #2 or 3 of the menstrual cycle.
3. BMI < 35.
4. No physical or gynecological abnormalities (including major uterine surgery) constituting a medical contraindication to embryo transfer and pregnancy including any known significant genetic disorders
5. Non-smoker for at least 3 months prior to study enrollment.
6. Normal antral follicle count (total ≥ 10).

Exclusion Criteria:

1. Greater than 1 previous miscarriage.
2. More than 1 previous failed IVF attempt.
3. Previous poor response to ovarian stimulation (peak E2 level <1,000 pg/ml or < 4 oocytes retrieved).
4. Presence of untreated hydrosalpinx.
5. Stage III or IV endometriosis.
6. Intent to have preimplantation genetic diagnosis (PGD) of embryos
7. Unwillingness to freeze or inseminate all eligible oocytes or embryos.
8. Male partner requiring surgical sperm retrieval (MESA or TESA).

Ages: 21 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Center for Advanced Reproductive Services patient population
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2009-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
oocyte survival | day of retrieval
fertilization | Day of retrieval
Embryo development | day 3 post retrieval

SECONDARY OUTCOMES:
Implantation | 3 weeks after transfer
Clinical pregnancy | 2 weeks after transfer
Miscarriage and live birth rates for those embryos derived from vitrified oocytes. | 9 months post transfer

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Benadiva, MD, HCLD, Principal Investigator — The Center for Advanced Reproductive Services, P.C.
Locations (1):
- The Center for Advanced Reproductive Services, Farmington, Connecticut, United States

REFERENCES:
- [Background] Antinori M, Licata E, Dani G, Cerusico F, Versaci C, Antinori S. Cryotop vitrification of human oocytes results in high survival rate and healthy deliveries. Reprod Biomed Online. 2007 Jan;14(1):72-9. doi: 10.1016/s1472-6483(10)60766-3. PMID 17207335
- [Background] Boldt J, Cline D, McLaughlin D. Human oocyte cryopreservation as an adjunct to IVF-embryo transfer cycles. Hum Reprod. 2003 Jun;18(6):1250-5. doi: 10.1093/humrep/deg242. PMID 12773454
- [Background] Cao YX, Xing Q, Li L, Cong L, Zhang ZG, Wei ZL, Zhou P. Comparison of survival and embryonic development in human oocytes cryopreserved by slow-freezing and vitrification. Fertil Steril. 2009 Oct;92(4):1306-1311. doi: 10.1016/j.fertnstert.2008.08.069. Epub 2008 Oct 18. PMID 18930218
- [Background] Carroll J, Depypere H, Matthews CD. Freeze-thaw-induced changes of the zona pellucida explains decreased rates of fertilization in frozen-thawed mouse oocytes. J Reprod Fertil. 1990 Nov;90(2):547-53. doi: 10.1530/jrf.0.0900547. PMID 2250252
- [Background] Chen C. Pregnancy after human oocyte cryopreservation. Lancet. 1986 Apr 19;1(8486):884-6. doi: 10.1016/s0140-6736(86)90989-x. PMID 2870356
- [Background] Chian RC, Huang JY, Tan SL, Lucena E, Saa A, Rojas A, Ruvalcaba Castellon LA, Garcia Amador MI, Montoya Sarmiento JE. Obstetric and perinatal outcome in 200 infants conceived from vitrified oocytes. Reprod Biomed Online. 2008 May;16(5):608-10. doi: 10.1016/s1472-6483(10)60471-3. PMID 18492361
- [Background] Ciotti PM, Porcu E, Notarangelo L, Magrini O, Bazzocchi A, Venturoli S. Meiotic spindle recovery is faster in vitrification of human oocytes compared to slow freezing. Fertil Steril. 2009 Jun;91(6):2399-407. doi: 10.1016/j.fertnstert.2008.03.013. Epub 2008 Aug 3. PMID 18675965
- [Background] Cobo A, Kuwayama M, Perez S, Ruiz A, Pellicer A, Remohi J. Comparison of concomitant outcome achieved with fresh and cryopreserved donor oocytes vitrified by the Cryotop method. Fertil Steril. 2008 Jun;89(6):1657-64. doi: 10.1016/j.fertnstert.2007.05.050. Epub 2007 Sep 24. PMID 17889865
- [Background] Fuku E, Xia L, Downey BR. Ultrastructural changes in bovine oocytes cryopreserved by vitrification. Cryobiology. 1995 Apr;32(2):139-56. doi: 10.1006/cryo.1995.1013. PMID 7743816
- [Background] Hong SW, Chung HM, Lim JM, Ko JJ, Yoon TK, Yee B, Cha KY. Improved human oocyte development after vitrification: a comparison of thawing methods. Fertil Steril. 1999 Jul;72(1):142-6. doi: 10.1016/s0015-0282(99)00199-5. PMID 10428163
- [Background] Kuwayama M, Vajta G, Kato O, Leibo SP. Highly efficient vitrification method for cryopreservation of human oocytes. Reprod Biomed Online. 2005 Sep;11(3):300-8. doi: 10.1016/s1472-6483(10)60837-1. PMID 16176668
- [Background] Kuleshova L, Gianaroli L, Magli C, Ferraretti A, Trounson A. Birth following vitrification of a small number of human oocytes: case report. Hum Reprod. 1999 Dec;14(12):3077-9. doi: 10.1093/humrep/14.12.3077. PMID 10601099
- [Background] Lucena E, Bernal DP, Lucena C, Rojas A, Moran A, Lucena A. Successful ongoing pregnancies after vitrification of oocytes. Fertil Steril. 2006 Jan;85(1):108-11. doi: 10.1016/j.fertnstert.2005.09.013. PMID 16412739
- [Background] Noyes N, Porcu E, Borini A. Over 900 oocyte cryopreservation babies born with no apparent increase in congenital anomalies. Reprod Biomed Online. 2009 Jun;18(6):769-76. doi: 10.1016/s1472-6483(10)60025-9. PMID 19490780